CLINICAL TRIAL: NCT06206902
Title: A Multicenter, Open Phase I Study to Evaluate the Safety and Pharmacokinetic Profile of F01 in Patients With Relapsed/Refractory Non-Hodgkin Lymphoma
Brief Title: F01 in the Treatment of Relapsed/Refractory Non-hodgkin's Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNC 103-CD19CAR NK-101
Record Dates: First submitted 2023-12-18; First posted 2024-01-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-12

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NK; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assigned Interventions (Experimental)
  Interventions: Drug: After preconditioning with chemotherapy, F01 will be evaluated.

INTERVENTIONS:
Drug: After preconditioning with chemotherapy, F01 will be evaluated. — Biological: 0.5-3×10^9 CAR+NK Cells, Treatment follows a lymphodepletion Drug: Fludarabine: 30 mg/m^2 (D-5~D-3) Drug: Cyclophosphamide: 300 mg/ m^2 (D-5~D-3)

SUMMARY:
This is a multicenter, open, Phase I clinical study to evaluate the safety and tolerability of F01 in subjects with relapsed/refractory non-Hodgkin lymphoma, and to determine MTD and/or RD.

DETAILED DESCRIPTION:
Approximately 55 participants with relapsed and/or refractory large B-cell lymphoma and follicular lymphoma stage 3b are planned to enroll. This study is divided into two stages: dose escalation and dose extension. In the phase of dose escalation, a single dose escalation study will be carried out first, and then multiple dose escalation studies will be carried out. In the dose expansion phase, up to 3 subjects who had previously received CD19-targeted CAR T cell therapy may enroll.

After the completion of the single dose escalation study, SRC will determine the MTD and/or RD of the single dose escalation phase based on the safety, pharmacokinetic profile (if applicable), immunogenicity, efficacy, and other data available at the time for each dose group. SRC will also determine whether the study will continue with multiple dose escalation studies or a single dose is sufficient to meet therapeutic needs. Multiple dose escalation can be skipped to provide recommendations for dose expansion phase studies based directly on single dose MTD and/or RD doses. After fully evaluating all opinions and data, the sponsor may choose to: 1) Multiple dose escalation studies are not conducted, and the MTD and/or RD doses with a single dose increase are directly entered into the dose expansion phase. In this case, enrolled subjects are continued to receive a single dose during the dose expansion phase to further confirm the safety and efficacy of subjects under RD dose; 2) After the single dose increment, enter the multi-dose increment study, and enter the dose extension phase after confirming the MTD and/or RD doses of multiple doses.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, gender unlimited.
2. ECOG score 0-2 points.
3. Large B-cell lymphoma or follicular lymphoma grade 3b was confirmed by histopathology.Large B-cell lymphomas include the following types as defined by WHO2016:

   * Diffuse large B lymphoma (DLBCL), non-specific type (NOS);
   * Large B-cell lymphoma rich in T cells/histiocytic cells;
   * EBV positive DLBCL, non-specific type (NOS);
   * Primary mediastinal (thymus) large B-cell lymphoma;
   * High-grade B-cell lymphoma, non-specific type (NOS) and high-grade B-cell lymphoma with MYC and BCL2 or BCL6 rearrangement;
   * Follicular lymphoma or other inert lymphoma transformed DLBCL.
4. Must have been previously treated with at least 2-line systemic anti-B-cell lymphoma. Participants must have received at least one course of anthracycline-based chemotherapy (except when absolutely contraindicated due to cardiac dysfunction) and at least one course of anti-CD20 immunotherapy (except in CD20-negative subjects or contraindicated due to severe toxicity).

   * Induction + consolidation + transplantation + maintenance treatment is a one-line system of treatment;
   * Anti-CD20 monotherapy does not count as 1-line systemic therapy;
   * Local radiotherapy does not count as 1-line systemic therapy.
5. Patients who have previously received targeted CD19 therapy (including monoclonal antibody, double antibody, CAR-T, experimental therapy, etc.) should provide histophistological reports during screening stage to confirm that CD19 expression is still present in lymphoma tissues after the last targeted CD19 therapy.
6. Imaging evidence indicates recurrent or refractory disease.

   * Definition of relapse: partial response (PR) or above achieved after the last treatment, with disease progression after treatment (except for those who meet the definition of refractory);
   * Refractory is defined as the failure to achieve a partial response (PR) or above from the last treatment, or relapse within 6 months after the last treatment regimen, or relapse within 12 months after autologous hematopoietic stem cell transplantation (ASCT). (If salvage therapy is performed after ASCT, subjects must have a response < PR to terminal therapy.).
7. According to Lugano 2014 lymphoma efficacy evaluation criteria (Cheson 2014), there is at least one measurable lesion (a measurable lesion is defined as a lymph node lesion with a diameter greater than 1.5cm and an extra-lymph node lesion with a diameter greater than 1.0cm).

   - Lesions that have previously received radiotherapy are only considered measurable if there is clear evidence of disease progression after completion of radiotherapy.
8. The expected survival is greater than 3 months.
9. Blood routine within 7 days from eluvial pre-treatment chemotherapy should meet the following requirements:

   * Absolute value of neutrophil (ANC) ≥ 1.0×109/L;
   * Hemoglobin (Hb) ≥ 80g/L;
   * Platelet count (PLT) ≥ 50×109/L.
10. Adequate liver, kidney, lung and heart function, defined as:

    1. Serum ALT and AST ≤ 2.5 times the upper limit of normal;
    2. Total bilirubin ≤ 1.5 times the upper limit of normal, except those with Gilbert syndrome, whose total bilirubin must ≤ 3.0 times the upper limit of normal;
    3. Creatinine clearance (estimated by Cockcroft Gault formula) (Appendix 2) ≥60ml/min;
    4. Under indoor ventilation conditions, the blood oxygen saturation in the non-oxygen state is ≥ 92%; There was no clinically significant pleural effusion;
    5. Left ventricular ejection fraction ≥ 50%; Echocardiography confirmed no clinically significant pericardial effusion. No clinically significant abnormalities were found in the ECG.
11. Subjects receiving hematopoietic growth factor support therapy, including erythropoietin (EPO), granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage-colony-stimulating factor (GM-CSF), and platelet agonist (TPO), There must be a 2-week interval between the last growth factor support treatment and the screening period evaluation; Screening platelet assessment should be at least 1 week away from the last platelet transfusion, and screening hemoglobin assessment should be at least 2 weeks away from the last red blood cell transfusion.
12. During the screening period, the serum pregnancy test results of fertile female subjects must be negative (women who have been surgically sterilized or have been menopausal for at least 2 years are considered not fertile). Fertile female subjects and male subjects must use highly effective contraceptive methods throughout the clinical study period and within 1 year after the last study treatment; At the same time, a commitment should be made not to donate eggs (egg cells, oocytes)/sperm for assisted reproduction within 1 year after the last study treatment.
13. Voluntarily participate in clinical trials and sign informed consent.

Exclusion Criteria:

1. Subjects with known allergic reactions, hypersensitivities, intolerances, or contraindications to F01 or any component of the drugs that may be used in the study, including fludarabine, cyclophosphamide, and tocilizumab, or who have previously experienced severe allergic reactions.
2. Primary central nervous system lymphoma.
3. Subjects with gastrointestinal lymphoma who had a history of ≥ grade 3 gastrointestinal bleeding in the 3 months prior to screening and those at risk of developing ≥ grade 3 gastrointestinal bleeding as assessed by investigators (CTCAE, version 5.0).
4. Subjects with a history of central nervous system lymphoma, lymphoma cells found in cerebrospinal fluid, and previous imaging findings of intracranial involvement of lymphoma could not be enrolled.
5. Performed allogeneic hematopoietic stem cell transplantation.
6. Autologous hematopoietic stem cell transplantation was performed within 3 months before eluvial pre-treatment chemotherapy.
7. Subjects who have previously received CD19-targeted CAR-NK therapy; The best efficacy of previous targeted CD19 CAR-T therapy < PR.
8. Major surgery or live vaccination within 28 days prior to screening.
9. Received the following anti-tumor therapy within the specified time frame before eluvial pre-treatment chemotherapy:

   1. Received small molecule targeted therapy within 3 weeks or 5 half-lives (whichever is longer);
   2. Receiving large molecule drug therapy within 4 weeks or 5 half-lives, whichever is longer (4 weeks for anti-CD20 antibody);
   3. Received cytotoxic therapy or modern Chinese medicine with anti-tumor effects within 3 weeks (liposomal adriamycin washout period was 4 weeks);
   4. Have received experimental therapy within 4 weeks (except for explicit placebo control);
   5. Received local palliative radiotherapy within 2 weeks.
10. At the time of screening, any aes associated with previous anti-lymphoma therapy have not returned to ≤ grade 1 or baseline (CTCAE version 5.0) (except for hair loss, blood routine and blood biochemical related AEs; Blood routine and blood biochemical test values refer to the inclusion criteria Article 9 and 10).
11. Previous CNS disease, such as seizures, cerebrovascular accidents (ischemia/bleeding), dementia, cerebellar disease, or any CNS related autoimmune disease.
12. At the time of screening, confirmed systemic autoimmune diseases requiring maintenance treatment or confirmed systemic autoimmune diseases were in the active phase.
13. Unstable cardiovascular function:

    1. Myocardial infarction occurred within 6 months prior to screening;
    2. Unstable angina occurred within 3 months prior to screening;
    3. Uncontrolled, clinically significant arrhythmias (e.g., persistent ventricular tachycardia, ventricular fibrillation, torsades de pointes arrhythmia );
    4. Mobitz II degree II or III degree atrioventricular block;
    5. New York Heart Function Society classification ≥3 congestive heart failure;
    6. Poorly controlled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg) or accompanied by hypertensive crisis or hypertensive encephalopathy;
14. Active hepatitis B virus (HBV), hepatitis C virus (HCV) infection at screening time. Admission of HBsAg positive and/or HBcAb positive but HBV-DNA negative, and/or HCVAb positive but HCV-RNA negative subjects (if the study center report includes a reference value range, the upper limit of normal HBV-DNA and HCV-RNA testing is based on the test values at each study center). Higher than the upper limit of the detection value is defined as "positive"; If the research center report only shows "negative/positive", "positive" is subject to the test report result).
15. Known serum HIV-positive or active HIV infection history, and syphilis screening antibody positive.
16. There is an active, uncontrolled infection that requires intravenous treatment with antibiotics, antiviral or antifungal agents within 14 days prior to eluvial pre-treatment chemotherapy; However, these drugs can be used for preventive treatment (including intravenous medication).
17. Malignant tumors that require treatment or have evidence of recurrence within 2 years prior to screening (except non-melanoma skin cancer that has been surgically removed, cured cervical carcinoma in situ, localized prostate cancer, low-stage bladder cancer, and ductal carcinoma in situ of the breast). However, subjects with tumors that had received >2 years of prior radical therapy and had no evidence of recurrence were admitted.
18. Use of drug combinations/combination therapies expressly prohibited by the protocol during screening.
19. The investigator believes that there is any life-threatening disease, medical condition, or organ system dysfunction that may affect the subject's safety or study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety of F01 cells | Up to 24 months
  The incidence, nature and severity of all adverse events, serious adverse events, and abnormal laboratory test results
Safety of F01 cells | Up to 1 month
  Incidence of DLT

SECONDARY OUTCOMES:
Response rate (ORR) of F01 cells | From 1 to 24 months after infusion
  Optimal objective response rate (ORR), 3-month ORR
Duration of response (DOR) of F01 cells | From 1 to 24 months after infusion
  Duration of response (DOR)
Progression-free survival (PFS) of F01 cells | From 1 to 24 months after infusion
  Progression-free survival (PFS)
Overall survival (OS) of F01 cells | From 1 to 24 months after infusion
  Overall survival (OS)
Maximum concentration of F01 cells | From 1 to 15 years after infusion or after learning of undetectable results
  Maximum concentration
Cmax of F01 cells | From 1 to 15 years after infusion or after learning of undetectable results
  Gene copy number amplification (Cmax)
Tmax of F01 cells | From 1 to 15 years after infusion or after learning of undetectable results
  Time to reach the maximum concentration (Tmax)
AUC0-last of F01 cells | From 1 to 15 years after infusion or after learning of undetectable results
  The area under the drug curve AUC0-last
Clast of F01 cells | From 1 to 15 years after infusion or after learning of undetectable results
  Last detectable concentration point (Clast)
Tlast of F01 cells | From 1 to 15 years after infusion or after learning of undetectable results
  Time of the last detectable concentration (Tlast)
Dynamic changes of cytokine levels | From 1 to 24 months
  The dynamic changes of cytokine levels in peripheral blood of subjects at baseline and after administration
Anti-CAR and IL-15 antibodies (ADA) | From 1 to 15 years after infusion or after learning of undetectable results
  The number of cases, positive rates, and duration of detection of anti-CAR and IL-15 antibodies (ADA) in subjects' serum at baseline and after administration
Peripheral blood lymphocyte subsets | From 1 to 24 months
  Dynamic changes of peripheral blood lymphocyte subsets compared with baseline after administration
Detection rate of replicable virus | From 1 to 15 years after infusion or after learning of undetectable results
  Detection rate of replicable virus

OTHER OUTCOMES:
The correlation among PK, PD, efficacy, and safety | From 1 to 24 months
  Explore the correlation among PK , PD（e.g. cytokines）, efficacy, and safety
The correlation among KIR mismatch , efficacy and safety | From 1 to 24 months
  Explore the correlation among KIR mismatch , efficacy and safety

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No